CLINICAL TRIAL: NCT00434278
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Pulmozyme Withdrawal on Exercise Tolerance in Cystic Fibrosis Subjects With Severe Lung Disease
Brief Title: A Trial of Pulmozyme Withdrawal on Exercise Tolerance in Cystic Fibrosis Subjects With Severe Lung Disease (TOPIC)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated for administrative reasons. There were no safety concerns.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z3877g
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis
Keywords: Lung disease; CF; Pulmozyme
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Dornase alfa (Experimental)
  Interventions: Drug: Dornase alfa

INTERVENTIONS:
Drug: Dornase alfa — 2.5 mg inhalation dose twice daily for 14±2 days
  Other Names: Pulmozyme
  Arms: Dornase alfa
Drug: placebo — 2.5 mg inhalation dose twice daily for 14±2 days
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled study of patients with severe, though stable, cystic fibrosis (CF) whose routine treatment included Pulmozyme. Patients were randomized to either continue Pulmozyme or have therapy withdrawn for 2 weeks (placebo group). Patients must have had stable CF symptoms without any change in therapy for 2 weeks prior to enrollment in order to participate.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form and, if applicable, Assent Form
* Age ≥ 14 years old at screening
* Proven diagnosis of CF
* Ability to perform acceptable and reproducible spirometry maneuvers at screening
* FVC ≤ 45% predicted for race, height, age, and sex at screening
* Chronic use of Pulmozyme for at least 3 months in the last year and daily or twice daily use during the 14 days prior to screening
* Stable regimen of chest physiotherapy (CPT) for at least 14 days prior to screening
* Ability to complete the 6-minute walk test at screening
* Ability to complete the 6-minute walk test and spirometry at Visit 2
* If on routine tobramycin solution for inhalation (i.e., TOBI®) or other cycled antibiotic therapy, intention to either start or stop therapy at the time of Visit 2 (based on routine therapy cycle; no other planned change in this antibiotic regimen for 28 days before or 28 days after Visit 2)
* Clinically stable with no change in medications during the 14 days prior to screening

Exclusion Criteria:

* Use of an investigational drug or device within 28 days prior to screening
* Previous episode of acute respiratory failure requiring assisted ventilation within 2 years prior to screening
* Previous lung transplant
* Any cardiac disease that would contraindicate performing the 6-minute walk test
* Pregnancy or nursing
* Known hypersensitivity or other contraindication to the use of Pulmozyme
* Previous completion or premature discontinuation of study drug or withdrawal from this study
* More than one prior screening failure for this study at any time or any prior screening failure for this study within the last 28 days

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Freemer, M.D., Study Director — Genentech, Inc.
Locations (40):
- United States (40):
  - University of Alabama, Birmingham, Alabama
  - Childrens Hospital of LA, Los Angeles, California
  - USC Adult CF Center, Los Angeles, California
  - CHOC, Orange, California
  - Capital Allergy Resp Dis Ctr, Sacramento, California
  - Ventura County Medical Ctr, Ventura, California
  - Nat'l Jewish Med/Research Ctr, Denver, Colorado
  - Pulm & Critical Care Assoc, Jacksonville, Florida
  - Univ of Miami, Miami, Florida
  - Central Florida Pulmonary Grou, Orlando, Florida
  - Brown Univ School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush Medical Center, Chicago, Illinois
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Univ of Michigan Hlth System, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Spectrum Hospital, Grand Rapids, Michigan
  - Michigan State University, Kalamazoo, Michigan
  - Univ of Minnesota Dept of Derm, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Pulmonary & Critical Care Med, St Louis, Missouri
  - Children's Lung Specialist, Las Vegas, Nevada
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - St. Peters Univ Hospital, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Long Island Jew Adult CF Ctr, New Hyde Park, New York
  - SUNY Upstate Medical Univ, Syracuse, New York
  - Duke Pediatric Clinical, Durham, North Carolina
  - Rainbow Babies & Child Hosp, Cleveland, Ohio
  - Toledo Childrens Hospital, Toledo, Ohio
  - Santiago Reyes MD-Private Prac, Oklahoma City, Oklahoma
  - CF Solutions, Inc, Tulsa, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical Univ of South Carolina, Charleston, South Carolina
  - Pediatric Pulmonary Assoc, Columbia, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Alamo Clinical Research Assoc, San Antonio, Texas
  - W Virginia Univ Health Sci Ctr, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; Dornase Alfa: 2.5 mg inhalation dose twice daily for 14±2 days (Visit 2 to Visit 3)
Period: Overall Study
Arm/Group | Placebo | Dornase Alfa
Started | 14 | 13
Completed | 12 | 13
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dornase Alfa | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (7.0) | 29.8 (10.0) | 27.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Distance Walked in the 6-minute Walk Test
Description: Change in distance walked was defined as (distance walked in 6 minutes at baseline [Day 0]) - (distance walked in 6 minutes at Day 14) in meters.
Time Frame: From baseline to Day 14
Population: Randomized patients. For placebo arm: 2 placebo patients who were randomized did not complete the study and therefore had no values to calculate change from baseline computation.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Placebo | Dornase Alfa
Number analyzed (Participants) | 12 | 13
Meters | 25.2 (79.8) | 26.9 (60.0)

2. Secondary Outcome: Change in Pulmonary Function as Measured by FEV1 and FVC
Description: FEV1 (forced expiratory volume in 1 second) and FVC (forced vital capacity) were recorded at Day 0 (baseline) and Day 14. Change in FEV1 and FVC from baseline to Day 14 was reported as a percentage of values predicted for age, height, and race.
Time Frame: From baseline to Day 14
Population: Randomized patients. Patients not included in this analysis did not meet ATS reproducibility criteria. Two patients in the placebo arm whose screening visit values did not meet ATS reproducibility criteria were randomized in error and completed the study.
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | Placebo | Dornase Alfa
Number analyzed (Participants) | 11 | 12
Percentage of predicted value
  FEV1 | -0.5 (4.1) | 0.2 (2.8)
  FVC | -1.2 (4.5) | 1.0 (4.8)

ADVERSE EVENTS:
Description: Randomized (same as safety-evaluable) patients. Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Placebo | Dornase Alfa
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/13
Other Adverse Events (participants affected / at risk) | 2/14 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Dornase Alfa (N=13)
Cystic Fibrosis (Congenital, familial and genetic disorders) | 1 | 1
Cystic Fibrosis Lung (Congenital, familial and genetic disorders) | 1 | 0
Distal Intestinal Obstruction Syndrome (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Dornase Alfa (N=13)
Cystic Fibrosis (Congenital, familial and genetic disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Because the study was terminated (for administrative reasons and infeasibility of enrollment), no conclusions can be made about the effect of Pulmozyme on exercise tolerance in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.